CLINICAL TRIAL: NCT02894320
Title: The Impact of Parkinson's Disease on Internal Preactivation of Sensory Effects of Intention-based Actions. A Subliminal Priming Study
Brief Title: Dynamic ASPECTS of Internal PRE-ACTIVATION of Effects Sensors of Voluntary ACTION in PARKINSON's Disease
Acronym: DYNIDEO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JBL_2014-28
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Voluntary action; Action-effect preactivation; Action-effect prediction
MeSH Terms: conditions — Parkinson Disease | interventions — Behavior Observation Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Parkinson's disease
  Interventions: Behavioral: Behavioral observation
- Healthy subjects: gender and age matched with Parkinson's disease patients, whose data will be extracted from an existing database
  Interventions: Behavioral: Behavioral observation

INTERVENTIONS:
Behavioral: Behavioral observation

SUMMARY:
The ability to predict sensory effects of people's own motor actions is a key component of Human action realization. Recent studies revealed this anticipation process to be involved in early and late stages of voluntary actions. Nevertheless, the question whether the action-effect anticipation is impacted or not by "motor pathologies", such as the Parkinson's disease, remains unclear. The current study is aimed to clarify this issue by using a subliminal priming paradigm in patients with Parkinson's disease and in matched control participants. Indeed, subliminal primes corresponding to visual action-effects are displayed at different time points before the actions' execution. Results should allow to determine whether or not the action-effect prediction is impaired at different stages of voluntary action in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years and older
* Parkinson's disease

Exclusion Criteria:

* Other pathology or neurological or psychiatric history
* Known pregnancy or breastfeeding
* Absence of affiliation to social security or universal health coverage (CMU)
* Person under legal protection
* Patient's opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Parkinson's disease, according to the MDS-UPDRS III (Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale), matched for gender and for age with healthy subjects from a database.
  This database has already been constituted by the CNRS (Centre national de la recherche scientifique, Laboratory of Psychology of Perception - UMR8242).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Reaction time | baseline
  time measured in seconds
error rate | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France